CLINICAL TRIAL: NCT03507647
Title: Mindfulness Based Cognitive Therapy for Bipolar Disorder
Acronym: MBCT-BD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Pro Persona Mental Health Care Foundation (Other); Altrecht (Other); Dimence (Unknown); PsyQ (Other)
Responsible Party: Principal Investigator, Anne Speckens, Prof. dr., Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBCT-BD-2017-2021
Record Dates: First submitted 2017-09-18; First posted 2018-04-25 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Bipolar Disorder
Keywords: randomized controlled trial; Mindfulness based cognitive therapy; clinical effectiveness; cost-effectiveness; working mechanisms
MeSH Terms: conditions — Bipolar Disorder | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, multicenter, prospective, evaluator-blinded clinical trial of MBCT added to treatment as usual (TAU) versus TAU alone
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed by independent research assistants blind to condition. Participants will be instructed to avoid unblinding as much as possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Cognitive Therapy added to usual care (Experimental): Patients in the MBCT arm will be invited to participate in MBCT added to their usual care.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy; Other: Usual Care
- Usual Care (Active Comparator): Usual care will typically consist of pharmacotherapy, psycho-education and self-management interventions (usually with a psychiatric nurse).
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — MBCT is a manualised group skills-training program (Segal, Williams & Teasdale 2012) consisting of eight weekly sessions of 2.5 hours, plus one day of silent practice. The program includes both formal and informal meditation exercises. Cognitive techniques that are part of the program are education, monitoring and scheduling of activities, identification of negative automatic thoughts and devising a relapse prevention plan.
  The MBCT treatment will be adapted to address the needs of patients with a bipolar disorder. A few examples of these adaptations are: (more) psychoeducation about manic symptoms in addition to the psychoeduction about depression; introducing the 3-minute breathing space earlier in the programme and more often during sessions, especially when strong emotions are present; repeatedly bringing the focus to self-care; and making use of the mindful movement (yoga) exercises more frequently.
  Other Names: MBCT; Mindfulness training
  Arms: Mindfulness Based Cognitive Therapy added to usual care
Other: Usual Care — Usual care will typically consist of pharmacotherapy, psycho-education and self-management interventions (usually with a psychiatric nurse). Usual care will not be restricted, except for proscribing high-frequency psychological interventions such as (group) cognitive behavioral therapy, for practical and methodological reasons.

SUMMARY:
The current study will be a randomized controlled trial (RCT) investigating the clinical and cost-effectiveness of Mindfulness-Based Cognitive Therapy (MBCT) as an adjunct to usual care, versus usual care alone, in reducing depressive symptoms in patients with bipolar disorder. Outcome measures include depressive, (hypo)manic and anxiety symptoms, risk of relapse/recurrence, functioning and mental health/well-being. The study also aims to explore possible working mechanisms such as improvements of mindfulness and self-compassion skills. The study will have a follow-up duration of 15 months from baseline.

DETAILED DESCRIPTION:
Introduction:

In the Netherlands, the lifetime prevalence of bipolar disorder (BD) is about 1.2% for men and 1.4% for women (de Graaf et al 2010). BD usually manifests itself during late adolescence or early adulthood. Its course is often chronic, with patients suffering from recurrent depressive, (hypo)manic, or mixed episodes, being symptomatic about half of the time (Judd 2002). Although hospital admissions are more common during manic episodes, illness-related disability is more strongly influenced by depressive episodes (Judd 2003). It has been estimated that about 25-50% of the patients with BD attempts suicide at least once and that the risk of suicide is about 5%(Hawton 2005).

Depressive symptoms in BD are common and have been associated with negative effects on the course of bipolar disorder in terms of functional impairment and quality of life (Gutiérrez-Rojas 2008). There are limited data on how to optimize the treatment of persistent or residual depressive symptoms in BD or to improve outcomes for those patients who do not benefit sufficiently from the available treatments. In addition, there is a need for interventions that not only target symptom reduction but also help patients to cope with their illness from a wider perspective, i.e. in terms of their personal values, goals, and social roles.

Mindfulness-Based Cognitive Therapy (MBCT) is an innovative intervention that has been shown effective in reducing depressive symptoms in unipolar recurrent depression (Aalderen 2012, Kuyken 2016) and appears promising for coping with severe mental illness (Davis and Kurzban 2012). Little is known about the effectiveness of MBCT for BD, with a number of pilot studies showing reductions in depressive symptoms, and one RCT showing reduction of anxiety symptoms. Considering the need for additional psychosocial treatments that not only target symptomatic but also personal recovery, these preliminary but encouraging findings warrant a larger RCT examining the efficacy of MBCT for BD in the Netherlands.

Aims:

As there are limited data on how to improve outcomes for those patients who do not benefit sufficiently from the available treatments, this study aims to compare MBCT to TAU as an adjunctive treatment to reduce depressive symptoms in patients with bipolar disorder. Outcomes of MBCT for BD patients will be examined both on a symptom level (depression, mania, anxiety, risk of relapse/recurrence) and in terms of functioning and mental health/well-being, including its possible working mechanisms such as improvements of mindfulness and self-compassion skills.

Method:

A randomized, multicenter, prospective, evaluator-blinded clinical trial of MBCT added to treatment as usual (TAU) versus TAU alone. Assessments will be conducted at baseline and at 3, 6, 9, 12 and 15 months follow-up.

The intervention will consist of usual care, and for half of the participants MBCT will be offered in adjunct. MBCT is a manualised group skills-training program (Segal, Williams & Teasdale 2012) designed as a relapse prevention programme for patients with recurrent depression. The training consists of eight weekly sessions of 2.5 hours, plus one day of silent practice. The program includes both formal and informal meditation exercises. Cognitive techniques that are part of the program are education, monitoring and scheduling of activities, identification of negative automatic thoughts and devising a relapse prevention plan.

The MBCT treatment will based on the 8-week MBCT course developed by Segal, Williams and Teasdale (2012), but will be adapted to address the needs of patients with a bipolar disorder. A few examples of these adaptations are: (more) psychoeducation about manic symptoms in addition to the psychoeducation about depression; introducing the 3-minute breathing space earlier in the programme and more often during sessions, especially when strong emotions are present; repeatedly bringing the focus to self-care; and making use of the mindful movement (yoga) exercises more frequently. All group sessions will be conducted at the respective mental health centres, with each group comprising 8-12 participants. MBCT courses will be taught by experienced and qualified mindfulness teachers, together with a health care professional specialised in the care for BD patients. Teacher competency will be assessed with the Mindfulness-Based Interventions - Teaching Assessment Criteria (Crane et al 2013), for which all trial sessions will be videotaped.

Usual care will consist of pharmacotherapy, psycho-education and self-management interventions (usually with a psychiatric nurse).

ELIGIBILITY:
Inclusion Criteria:

* bipolar I or II disorder
* having suffered at least two lifetime depressive episodes, either current or in (partial) remission at baseline (according to SCID assessment)
* Young Mania Rating Scale score < 8

Exclusion Criteria:

* a manic episode in the 3 months before the start of the trial
* lifetime diagnosis of schizophrenia or schizoaffective disorder, current substance abuse disorder, organic brain syndrome, antisocial or borderline personality disorder
* risk of suicide or aggression
* the presence of a concurrent significant medical condition impeding the ability to participate
* currently receiving regular psychological therapy
* previous participation in a MBCT or MBSR course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Inventory of Depressive Symptomatology | Change between baseline and 3 months
  A clinican-administered interview assessing the severity of depressive symptoms

SECONDARY OUTCOMES:
Structured Clinical Interview for DSM-IV-TR Disorders | Change between baseline and 15 months
  Diagnostic instrument to assess relapse of depressive or (hypo)manic episode
Young Mania Rating Scale | Change between baseline and 3 months
  Young Mania Rating Scale (YMRS) Dutch translation. The YMRS is an 11-item clinician-administered rating scale to assess the severity of (hypo)manic symptoms. It was found to be a reliable, valid, and sensitive rating scale to measure the severity of mania (Young et al., 1978). Its total score ranges from 0 (no (hypo)manic symptoms) to 44 (severe manic symptoms).
Young Mania Rating Scale | Change between baseline and 15 months
  Young Mania Rating Scale (YMRS) Dutch translation. The YMRS is an 11-item clinician-administered rating scale to assess the severity of (hypo)manic symptoms. It was found to be a reliable, valid, and sensitive rating scale to measure the severity of mania (Young et al., 1978). Its total score ranges from 0 (no (hypo)manic symptoms) to 44 (severe manic symptoms).
Functioning Assessment Short Test | Change between baseline and 3 months
  Brief instrument designed to assess the main functioning problems experienced by psychiatric patients, particularly bipolar patients
Functioning Assessment Short Test | Change between baseline and 15 months
  Brief instrument designed to assess the main functioning problems experienced by psychiatric patients, particularly bipolar patients
State/Trait Anxiety Inventory | Change between baseline and 3 months
  self-report measure for assessing both state and trait levels of anxiety
State/Trait Anxiety Inventory | Change between baseline and 15 months
  self-report measure for assessing both state and trait levels of anxiety
Ruminative Response Scale - brooding subscale | Change between baseline and 3 months
  Brooding subscale of the extended version of the Ruminative Response Scale (RRS-EXT). The authors reported adequate internal consistency (α = .79) and test-retest stability (α = .62, with a one year time interval) for the brooding subscale, which consists of five items. We select the brooding subscale because over time, brooding, or rumination, has been more strongly related to levels of depression (Treynor et al., 2003). Items are scored between 1 ((almost) never) to 4 ((almost) always and subscale score ranges between 5 and 20. A higher score indicates a higher level of ruminative brooding.
Ruminative Response Scale - brooding subscale | Change between baseline and 15 months
  Brooding subscale of the extended version of the Ruminative Response Scale (RRS-EXT). The authors reported adequate internal consistency (α = .79) and test-retest stability (α = .62, with a one year time interval) for the brooding subscale, which consists of five items. We select the brooding subscale because over time, brooding, or rumination, has been more strongly related to levels of depression (Treynor et al., 2003). Items are scored between 1 ((almost) never) to 4 ((almost) always and subscale score ranges between 5 and 20. A higher score indicates a higher level of ruminative brooding.
Five Facet Mindfulness Questionnaire, short form | Change between baseline and 3 months
  Self-report measure consisting of 24 items divided into the subscales observing, describing, acting with awareness, non-judging and non-reactivity.
Five Facet Mindfulness Questionnaire, short form | Change between baseline and 15 months
  Self-report measure consisting of 24 items divided into the subscales observing, describing, acting with awareness, non-judging and non-reactivity.
Self-Compassion Scale | Change between baseline and 3 months
  Self-Compassion Scale - short form (SCS-SF). The present study will use the 12-item Dutch short-form version of the SCS-SF to measure self-compassion. The scale consists of six components, including self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification. The SCS-SF has good reliability and validity (Raes et al., 2011). In the short form, each scale consists of 2 items scored between 1 ((almost) never) to 7 ((almost) always) and subscale score ranges between 2 and 14. A higher score indicates a higher level of self-kindness, common humanity, and mindfulness, and lower scores of self-judgment, isolation, and over-identification. Total scores range from 12 to 84 (summed subscale scores), a higher score indicates a higher level of selfcompassion.
Self-Compassion Scale | Change between baseline and 15 months
  Self-Compassion Scale - short form (SCS-SF). The present study will use the 12-item Dutch short-form version of the SCS-SF to measure self-compassion. The scale consists of six components, including self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification. The SCS-SF has good reliability and validity (Raes et al., 2011). In the short form, each scale consists of 2 items scored between 1 ((almost) never) to 7 ((almost) always) and subscale score ranges between 2 and 14. A higher score indicates a higher level of self-kindness, common humanity, and mindfulness, and lower scores of self-judgment, isolation, and over-identification. Total scores range from 12 to 84 (summed subscale scores), a higher score indicates a higher level of selfcompassion.
Mental Health Continuum - short form | Change between baseline and 3 months
  A 14-item self-report questionnaire that assesses emotional, psychological and social well-being
Mental Health Continuum - short form | Change between baseline and 15 months
  A 14-item self-report questionnaire that assesses emotional, psychological and social well-being
Inventory of Depressive Symptomatology | 6 months
  A clinican-administered interview assessing the severity of depressive symptoms
Inventory of Depressive Symptomatology | 9 months
  A clinican-administered interview assessing the severity of depressive symptoms
Inventory of Depressive Symptomatology | 12 months
  A clinican-administered interview assessing the severity of depressive symptoms
Inventory of Depressive Symptomatology | 15 months
  A clinican-administered interview assessing the severity of depressive symptoms

OTHER OUTCOMES:
Euro-Quality of Life 5D-5L | baseline
  Short self-report instrument to assess quality adjusted life years
Euro-Quality of Life 5D-5L | 3 months
  Short self-report instrument to assess quality adjusted life years
Euro-Quality of Life 5D-5L | 6 months
  Short self-report instrument to assess quality adjusted life years
Euro-Quality of Life 5D-5L | 9 months
  Short self-report instrument to assess quality adjusted life years
Euro-Quality of Life 5D-5L | 12 months
  Short self-report instrument to assess quality adjusted life years
Euro-Quality of Life 5D-5L | 15 months
  Short self-report instrument to assess quality adjusted life years
Trimbos/iMTA Questionnaire on Costs associated with Psychiatric illness | baseline
  Health service receipt interview designed for economic evaluations in the Netherlands
Trimbos/iMTA Questionnaire on Costs associated with Psychiatric illness | 3 months
  Health service receipt interview designed for economic evaluations in the Netherlands
Trimbos/iMTA Questionnaire on Costs associated with Psychiatric illness | 6 months
  Health service receipt interview designed for economic evaluations in the Netherlands
Trimbos/iMTA Questionnaire on Costs associated with Psychiatric illness | 9 months
  Health service receipt interview designed for economic evaluations in the Netherlands
Trimbos/iMTA Questionnaire on Costs associated with Psychiatric illness | 12 months
  Health service receipt interview designed for economic evaluations in the Netherlands
Trimbos/iMTA Questionnaire on Costs associated with Psychiatric illness | 15 months
  Health service receipt interview designed for economic evaluations in the Netherlands

CONTACTS AND LOCATIONS:
Overall Officials: Anne Speckens, Prof., Principal Investigator — Radboud University Medical Center
Locations (4):
- Netherlands (4):
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - Dimence GGZ, Deventer
  - Pro Persona, Nijmegen
  - Altrecht GGZ, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
The authors intend to make the data available to other researchers after completion of the study and will comply with open access procedures, including open access publishing, as much as possible.

REFERENCES:
- [Derived] Hanssen I, Huijbers M, Regeer E, Lochmann van Bennekom M, Stevens A, van Dijk P, Boere E, Havermans R, Hoenders R, Kupka R, Speckens AE. Mindfulness-based cognitive therapy v. treatment as usual in people with bipolar disorder: A multicentre, randomised controlled trial. Psychol Med. 2023 Oct;53(14):6678-6690. doi: 10.1017/S0033291723000090. Epub 2023 Mar 7. PMID 39625263
- [Derived] Hanssen I, Scheepbouwer V, Huijbers M, Regeer E, Lochmann van Bennekom M, Kupka R, Speckens A. Adverse or therapeutic? A mixed-methods study investigating adverse effects of Mindfulness-Based Cognitive Therapy in bipolar disorder. PLoS One. 2021 Nov 4;16(11):e0259167. doi: 10.1371/journal.pone.0259167. eCollection 2021. PMID 34735517
- [Derived] Hanssen I, van der Horst N, Boele M, Lochmann van Bennekom M, Regeer E, Speckens A. The feasibility of mindfulness-based cognitive therapy for people with bipolar disorder: a qualitative study. Int J Bipolar Disord. 2020 Nov 11;8(1):33. doi: 10.1186/s40345-020-00197-y. PMID 33175338
- [Derived] Hanssen I, Huijbers MJ, Lochmann-van Bennekom MWH, Regeer EJ, Stevens AWMM, Evers SMAA, Wensing M, Kupka RW, Speckens AEM. Study protocol of a multicenter randomized controlled trial of mindfulness-based cognitive therapy and treatment as usual in bipolar disorder. BMC Psychiatry. 2019 Apr 30;19(1):130. doi: 10.1186/s12888-019-2115-6. PMID 31039765

DOCUMENTS (1):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT03507647/Prot_000.pdf